CLINICAL TRIAL: NCT03281265
Title: A Retrospective Multicenter Study of HBV-related Pre-acute-on-chronic Liver Failure in China
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-07

CONDITIONS: Liver Failure, Acute on Chronic; Liver Injury
Keywords: pre-acute-on-chronic liver failure; hepatitis B
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard treatment

SUMMARY:
The definition and diagnostic criteria of Acute-on-chronic liver failure (ACLF) has been well established by EASL CANONIC study. However, patients with high risk to develop ACLF has not been determined, yet. The aim of current study is to establish a preliminary pre-ACLF definition, and to demonstrate the corresponding risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis B virus infection;
2. Any of the followings: Alanine aminotransferase (ALT)≥3 upper limit of laboratory reference (ULN); Aspartate aminotransferase (AST)≥3 ULN; Serum bilirubin≥2 ULN; Acute decompensation (ascites, hepatic encephalopathy, variceal hemorrhage and/or bacterial infections)

Exclusion Criteria:

1. Previous decompensation;
2. those who had hepatocellular carcinoma or other types of malignancies;
3. those who combined with severe chronic extra-hepatic disease;
4. pregnant;
5. received liver transplantation or kidney transplantation before or after admission;
6. readmission;
7. death within 24 hours.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with HBV-related compensated liver disease and acute liver injury or decompensation.
Sampling Method: Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
28-day ACLF progression | 28-day
  progressed to EASL defined ACLF
28-day mortality | 28-day
  death within 28-day

SECONDARY OUTCOMES:
90-day mortality | 90-day
  death within 90-day

IPD SHARING:
Plan to Share IPD: Undecided